CLINICAL TRIAL: NCT01984684
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Controlled Study to Evaluate the Efficacy + Safety of IV + Oral Delafloxacin Compared With Vancomycin + Aztreonam in Patients With Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Brief Title: Delafloxacin vs Vancomycin and Aztreonam for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RX-3341-303
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections; Skin Structures and Soft Tissue Infections
Keywords: Bacterial skin infection; infection; skin; delafloxacin; vancomycin; aztreonam; methicillin-resistant Staphylococcus aureus (MRSA) bacteria; bacterial infection; Anti-Infective Agents
MeSH Terms: conditions — Soft Tissue Infections; Skin Diseases, Bacterial; Infections; Bacterial Infections | interventions — delafloxacin; Vancomycin; Aztreonam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delafloxacin (Experimental): Delafloxacin 300 mg IV Q12H for 6 doses, then Delafloxacin 450 mg oral tablet Q12H for a minimum of 10 up to a maximum of 28 doses total
  Interventions: Drug: delafloxacin
- Vancomycin plus Aztreonam (Active Comparator): Vancomycin 15 mg/kg IV plus two grams Aztreonam every 12 hours for a minimum of 10 up to a maximum of 28 doses total (Aztreonam was discontinued as soon as possible if a gram-negative organism was not identified in baseline cultures)
  Interventions: Drug: vancomycin; Drug: aztreonam

INTERVENTIONS:
Drug: delafloxacin
  Other Names: RX-3341
  Arms: Delafloxacin
Drug: vancomycin
  Arms: Vancomycin plus Aztreonam
Drug: aztreonam
  Arms: Vancomycin plus Aztreonam

SUMMARY:
The purpose of this study is to evaluate the effects of Delafloxacin versus Vancomycin plus Aztreonam in the treatment of patients with acute bacterial skin and soft tissue infections.

DETAILED DESCRIPTION:
The purpose of this study is to determine if delafloxacin, an investigational drug, is safe and effective in the treatment of skin and nearby tissue infections compared with a combination of other antibiotics, vancomycin and aztreonam.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) men or women with a diagnosis of ABSSSI (cellulitis/erysipelas, wound infection, major cutaneous abscess, or burn infection) with surrounding redness of a minimum surface area of 75 cm^2 and at least two signs of systemic infection
* In the opinion of the investigator, the subject must require and be a suitable candidate for IV antibiotic therapy, and the subject must be able and willing to comply with protocol requirements

Exclusion Criteria:

* A medical history of significant hypersensitivity or allergic reaction to quinolones, beta-lactams, vancomycin, or vancomycin derivatives according to the judgment of the investigator.
* Women who are pregnant or lactating.
* Any chronic or underlying skin condition at the site of infection that may complicate the assessment of response, including infection involving a prosthetic joint, human or animal bite, osteomyelitis, decubitus ulcer, diabetic foot ulcer, septic arthritis, mediastinitis, necrotizing fasciitis, anaerobic cellulitis, or synergistic necrotizing cellulitis, myositis, tendinitis, endocarditis, sustained shock, gangrene or gas gangrene; burns covering ≥10% of body surface area; severely compromised immune system, severely impaired arterial blood supply to an extremity with an ABSSSI, deep vein thrombosis or superficial thrombophlebitis, and requiring either an amputation or multiple debridement procedures.
* Receipt of systemic antibiotic therapy in the 14 days before enrollment unless 1 of the following was documented:

  * Received ≥ 48 hours of antibiotic therapy for ABSSSI AND clinical progression is documented (i.e., not by patient history alone).
  * Recently (within 14 days) completed a treatment course with an antibacterial drug for an infection other than ABSSSI and the drug does not have activity against bacterial pathogens that cause ABSSSI.
  * Received only 1 dose of either a single, potentially effective, short-acting antimicrobial drug or drug regimen for ABSSSI.
* Any underlying disease that, in the opinion of the investigator, could interfere with the subject's ability to participate in the study including severe cardiac disease, known history of liver disease, end-stage renal disease, malignancy, psychiatric disorder, ongoing treatment for seizures or untreated history of seizures, or life expectancy of < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue K Cammarata, MD, Study Director — Melinta Therapeutics, Inc.
Locations (94):
- United States (31):
  - Melinta 303 Study Site, Mobile, Alabama
  - Melinta 303 Study Site, Montgomery, Alabama
  - Melinta 303 Study Site, Anaheim, California
  - Melinta 303 Study Site, Chula Vista, California
  - Melinta 303 Study Site, La Mesa, California
  - Melinta 303 Study Site, Long Beach, California
  - Melinta 303 Study Site, Modesto, California
  - Melinta 303 Study Site, Oceanside, California
  - Melinta 303 Study Site, San Diego, California
  - Melinta 303 Study Site, Stockton, California
  - Melinta 303 Study Site, Torrance, California
  - Melinta 303 Study Site, DeLand, Florida
  - Melinta 303 Study Site, Orlando, Florida
  - Melinta 303 Study Site, Columbus, Georgia
  - Melinta 303 Study Site, Savannah, Georgia
  - Melinta 303 Study Site, Eunice, Louisiana
  - Melinta 303 Study Site, Springfield, Massachusetts
  - Melinta 303 Study Site, Minneapolis, Minnesota
  - Melinta 303 Study Site, Butte, Montana
  - Melinta 303 Study Site, Lincoln, Nebraska
  - Melinta 303 Study Site, Las Vegas, Nevada
  - Melinta 303 Study Site, Somers Point, New Jersey
  - Melinta 303 Study Site, Teaneck, New Jersey
  - Melinta 303 Study Site, Columbus, Ohio
  - Melinta 303 Study Site, Toledo, Ohio
  - Melinta 303 Study Site, Rapid City, South Dakota
  - Melinta 303 Study Site, Jackson, Tennessee
  - Melinta 303 Study Site, Smyrna, Tennessee
  - Melinta 303 Study Site, Channelview, Texas
  - Melinta 303 Study Site, Houston, Texas
  - Melinta 303 Study Site, San Antonio, Texas
- Argentina (4):
  - Melinta 303 Study Site, La Plata, Buenos Aires
  - Melinta 303 Study Site, Rosario, Santa Fe Province
  - Melinta 303 Study Site, Córdoba
  - Melinta 303 Study Site, Santa Fe
- Brazil (7):
  - Melinta 303 Study Site, Salvador, Estado de Bahia
  - Melinta 303 Study Site, Belo Horizonte, Minas Gerais
  - Melinta 303 Study Site, Lavras, Minas Gerais
  - Melinta 303 Study Site, Passo Fundo, Rio Grande do Sul
  - Melinta 303 Study Site, Campinas, São Paulo
  - Melinta 303 Study Site, São José do Rio Preto, São Paulo
  - Melinta 303 Study Site, São Paulo
- Bulgaria (5):
  - Melinta 303 Study Site, Pleven
  - Melinta 303 Study Site, Plovdiv
  - Melinta 303 Study Site, Rousse
  - Melinta 303 Study Site, Sofia
  - Melinta 303 Study Site, Varna
- Chile (2):
  - Melinta 303 Study Site, Santiago
  - Melinta 303 Study Site, Temuco
- Estonia (4):
  - Melinta 303 Study Site, Kohtla-Järve
  - Melinta 303 Study Site, Tallinn
  - Melinta 303 Study Site, Tartu
  - Melinta 303 Study Site, Võru
- Georgia (4):
  - Melinta 303 Study Site, Batumi
  - Melinta 303 Study Site, Kutaisi
  - Melinta 303 Study Site, Tbilisi
  - Melinta 303 Study Site, Zugdidi
- Hungary (5):
  - Melinta 303 Study Site, Kaposvár
  - Melinta 303 Study Site, Kecskemét
  - Melinta 303 Study Site, Nyíregyháza
  - Melinta 303 Study Site, Szeged
  - Melinta 303 Study Site, Veszprém
- Latvia (4):
  - Melinta 303 Study Site, Daugavpils
  - Melinta 303 Study Site, Liepāja
  - Melinta 303 Study Site, Rēzekne
  - Melinta 303 Study Site, Riga
- Mexico (2):
  - Melinta 303 Study Site, Guadalajara, Jalisco
  - Melinta 303 Study Site, Monterrey, Nuevo León
- Melinta 303 Study Site, Chisinau, Moldova
- Peru (4):
  - Melinta 303 Study Site, Trujillo, La Libertad
  - Melinta 303 Study Site, Cusco
  - Melinta 303 Study Site, Lima
  - Melinta 303 Study Site, Loreto
- Romania (5):
  - Melinta 303 Study Site, Cluj-Napoca, Cluj
  - Melinta 303 Study Site, Craiova, Dolj
  - Melinta 303 Study Site, Timișoara, Timiș County
  - Melinta 303 Study Site, Bucharest
  - Melinta 303 Study Site, Târgu Mureş
- Slovakia (2):
  - Melinta 303 Study Site, Banská Bystrica
  - Melinta 303 Study Site, Prešov
- South Korea (8):
  - Melinta 303 Study Site, Wŏnju, Gang'weondo
  - Melinta 303 Study Site, Ansan, Gyeonggido
  - Melinta 303 Study Site, Goyang, Gyeonggido
  - Melinta 303 Study Site, Daegu
  - Melinta 303 Study Site, Daejeon
  - Melinta 303 Study Site, Gwangju
  - Melinta 303 Study Site, Incheon
  - Melinta 303 Study Site, Seoul
- Taiwan (6):
  - Melinta 303 Study Site, Kaohsiung City
  - Melinta 303 Study Site, New Taipei City
  - Melinta 303 Study Site, Taichung
  - Melinta 303 Study Site, Tainan
  - Melinta 303 Study Site, Taipei
  - Melinta 303 Study Site, Zhonghe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lodise T, Corey R, Hooper D, Cammarata S. Safety of Delafloxacin: Focus on Adverse Events of Special Interest. Open Forum Infect Dis. 2018 Sep 10;5(10):ofy220. doi: 10.1093/ofid/ofy220. eCollection 2018 Oct. PMID 30349845
- [Derived] O'Riordan W, McManus A, Teras J, Poromanski I, Cruz-Saldariagga M, Quintas M, Lawrence L, Liang S, Cammarata S; PROCEED Study Group. A Comparison of the Efficacy and Safety of Intravenous Followed by Oral Delafloxacin With Vancomycin Plus Aztreonam for the Treatment of Acute Bacterial Skin and Skin Structure Infections: A Phase 3, Multinational, Double-Blind, Randomized Study. Clin Infect Dis. 2018 Aug 16;67(5):657-666. doi: 10.1093/cid/ciy165. PMID 29518178
- [Derived] McCurdy S, Lawrence L, Quintas M, Woosley L, Flamm R, Tseng C, Cammarata S. In Vitro Activity of Delafloxacin and Microbiological Response against Fluoroquinolone-Susceptible and Nonsusceptible Staphylococcus aureus Isolates from Two Phase 3 Studies of Acute Bacterial Skin and Skin Structure Infections. Antimicrob Agents Chemother. 2017 Aug 24;61(9):e00772-17. doi: 10.1128/AAC.00772-17. Print 2017 Sep. PMID 28630189

RESULTS

PARTICIPANT FLOW:
Groups:
- Delafloxacin: 300 mg IV Q12H for 6 doses, 450 mg oral tablet Q12H for a minimum of 10 up to a maximum of 28 doses total
- Vancomycin Plus Aztreonam: Vancomycin 15 mg/kg IV plus two grams Aztreonam every 12 hours for a minimum of 10 up to a maximum of 28 doses total
Period: Overall Study
Arm/Group | Delafloxacin | Vancomycin Plus Aztreonam
Started | 423 | 427
Completed | 366 | 368
Not Completed | 57 | 59
Not completed — Lost to Follow-up | 25 | 24
Not completed — Adverse Event | 8 | 12
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Lack of Efficacy | 3 | 6
Not completed — Physician Decision | 4 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Death | 0 | 1
Not completed — Noncompliance with study drug | 2 | 1
Not completed — Subject incarcerated | 1 | 0
Not completed — Study drug not available at site | 1 | 1
Not completed — Subject had inadequate IV access | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all patients who were randomly assigned to treatment.
Groups:
- Delafloxacin: 300mg iv Q12H for 6 doses, 450mg oral tablet Q12H for a minimum of 10 up to a maximum of 28 doses total
- Vancomycin Plus Aztreonam: Vancomycin 15mg/kg iv plus two grams Aztreonam every 12 hours for a minimum of 10 up to a maximum of 28 doses total
- Total: Total of all reporting groups
Arm/Group | Delafloxacin | Vancomycin Plus Aztreonam | Total
Number analyzed (Participants) | 423 | 427 | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (15.98) | 50.2 (16.03) | 50.7 (16.00)
Age, Customized [Count of Participants; unit: Participants]
  <= 65 years | 344 | 352 | 696
  > 65 years | 79 | 75 | 154
  > 75 years | 35 | 31 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 151 | 312
  Male | 262 | 276 | 538
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 132 | 99 | 231
  Not Hispanic or Latino | 291 | 328 | 619
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 7 | 19
  Asian | 11 | 15 | 26
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 13 | 18 | 31
  White | 348 | 355 | 703
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 37 | 30 | 67
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 165 | 173 | 338
  North America | 202 | 196 | 398
  Mexico | 8 | 4 | 12
  Brazil | 0 | 5 | 5
  Chile | 1 | 1 | 2
  Peru | 34 | 29 | 63
  South Korea | 8 | 13 | 21
  Taiwan | 1 | 1 | 2
  Argentina | 4 | 5 | 9
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m2] | 30.4 (7.44) | 30.7 (7.54) | 30.5 (7.49)
BMI category [Count of Participants; unit: Participants]
  < 30 kg/m2 | 212 | 213 | 425
  >= 30 kg/m2 | 211 | 214 | 425
Presence of diabetes [Count of Participants; unit: Participants] | 53 | 54 | 107

OUTCOME MEASURES:

1. Primary Outcome: Objective Response of ≥20% Reduction in Lesion Erythema Area Compared to Baseline at 48 to 72 Hours After Initiation of Treatment as Determined by Digital Measurements of the Leading Edge.
Description: A patient was considered a responder if s/he had a ≥20% reduction in size of the area of erythema associated with the baseline ABSSSI, as determined by digital planimetry of the leading edge and had none of the reasons for clinical failure; a patient was considered a non-responder (failure) if s/he had <20% reduction in size of the area of erythema associated with the baseline ABSSSI as determined by digital planimetry of the leading edge, or had major intervention such as another antibiotic or surgical intervention or died within 74 hours after initiation of study drug.
Time Frame: 48 to 72 hrs after starting treatment
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Vancomycin Plus Aztreonam
Number analyzed (Participants) | 423 | 427
Participants
  Responder | 354 | 344
  Nonresponder | 69 | 83
Statistical Analysis 1: Comparison: Delafloxacin vs Vancomycin Plus Aztreonam; Test type: Non-Inferiority — A 2-sided 95% confidence interval (CI) for noninferiority testing was computed based on the difference in responder rates for vancomycin + aztreonam and delafloxacin at the primary endpoint. If the upper limit (UL) of the CI was less than 0.10, delafloxacin would be considered noninferior to vancomycin + aztreonam; Difference in Responder Rates = 3.1, 95% CI 2-sided [-2.0 to 8.3]

2. Secondary Outcome: Investigator-assessed Response of Signs and Symptoms of Infection at the Follow up Visit (European Medicines Agency [EMA] Primary Endpoint)
Description: A patient was considered a Cure if all baseline signs and symptoms of ABSSSI had resolved; if some symptoms remained, but the patient was improved to the extent that no additional antibiotic treatment was necessary, the response was Improved. A patient was considered a Failure for any of the following reasons: nonstudy antibacterial drug therapy was required because of lack of efficacy after at least 4 doses of study drug or for a treatment-related AE; study antibacterial drug therapy was required for longer than 28 doses; and/or unplanned surgical intervention was needed after study entry except for limited bedside debridement and standard wound care. Improved and Indeterminate responses were considered failures in the primary analysis.
  A sensitivity analysis was also performed, in which the assigned responses were Success (Cure + Improved) or Failure (Failure + Indeterminate/Missing).
Time Frame: Study Day 14 ± 1
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Vancomycin Plus Aztreonam
Number analyzed (Participants) | 423 | 427
Participants
  Cure | 244 | 255
  Improved | 125 | 107
  Failure | 17 | 21
  Indeterminate/Missing | 37 | 44
Statistical Analysis 1: Comparison: Delafloxacin vs Vancomycin Plus Aztreonam; Test type: Non-Inferiority — Analysis of the investigator's assessment of response of signs and symptoms of infection (cure only) was performed using the Miettinen-Nurminen method without stratification for the ITT analysis set; Difference in Cure Rates = -2.0, 95% CI 2-sided [-8.6 to 4.6]

3. Secondary Outcome: Investigator-assessed Response of Signs and Symptoms of Infection at the Late Follow-up Visit
Description: as for outcome 2
Time Frame: Study Day 21 to 28
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Vancomycin Plus Aztreonam
Number analyzed (Participants) | 423 | 427
Participants
  Cure | 287 | 303
  Improved | 66 | 48
  Failure | 21 | 24
  Indeterminate/Missing | 49 | 52
Statistical Analysis 1: Comparison: Delafloxacin vs Vancomycin Plus Aztreonam; Test type: Non-Inferiority — Analysis of the investigator's assessment of response (cure only) at the Late Follow-up Visit was assessed using the Miettinen-Nurminen method without stratification; Difference in Cure Rates = -3.1, 95% CI 2-sided [-9.3 to 3.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the patient signed informed consent through the follow-up telephone contact 30 (+3) days after the last dose of study drug (up to 48 days).
Description: AE data are only included for the safety population which included all patients in the ITT population who received at least 1 dose of study drug.
Arm/Group | Delafloxacin | Vancomycin Plus Aztreonam
All-Cause Mortality (participants affected / at risk) | 0/417 | 2/425
Serious Adverse Events (participants affected / at risk) | 16/417 | 17/425
Other Adverse Events (participants affected / at risk) | 55/417 | 32/425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delafloxacin (N=417) | Vancomycin Plus Aztreonam (N=425)
Myocardial infarction (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Intestinal ischemia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Systemic inflammatory response symdrome (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 3
Erysipelas (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 4 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2
ALT increased (Investigations) | 1 | 0
AST increased (Investigations) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of the colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delafloxacin (N=417) | Vancomycin Plus Aztreonam (N=425)
Diarrhea (Gastrointestinal disorders) | 32 | 14
Nausea (Gastrointestinal disorders) | 32 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Melinta has the right to first publication of results, which would be made in conjunction with the PIs from all appropriate sites. Thereafter, PIs may publish results provided the PI submits the proposed publication to Melinta for review at least 60 days prior to the date of the proposed publication. Melinta may remove any information that is considered confidential and/or proprietary. If a publication is not submitted within 12 months of study conclusion, the PI may publish results.